CLINICAL TRIAL: NCT00800215
Title: A Multicenter, Double-blind, Double-dummy, Randomized Trial to Investigate the Safety, Tolerability and Pharmacokinetics of Intravenous SPM 927 as Replacement for Oral SPM 927 in Subjects With Partial Seizures With or Without Secondary Generalization
Brief Title: A Trial to Investigate the Safety, Tolerability and Pharmacokinetics of Intravenous SPM 927
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: UCB Pharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SP616
Record Dates: First submitted 2008-12-01; First posted 2008-12-02 (Estimated); Last update posted 2024-04-19 (Actual); Status verified 2024-04

CONDITIONS: Epilepsy
Keywords: Epilepsy
MeSH Terms: conditions — Epilepsy | interventions — 2-(acetylamino)-3-methoxy-N-(phenylmethyl)-, (2R)-; Lacosamide

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- 1 (Experimental)
  Interventions: Drug: iv SPM 927 and oral placebo tablet
- 2 (Placebo Comparator)
  Interventions: Drug: oral SPM 927 tablet and iv placebo
- 3 (Experimental)
  Interventions: Drug: iv SPM 927 and oral placebo tablet
- 4 (Placebo Comparator)
  Interventions: Drug: oral SPM 927 tablet and iv placebo

INTERVENTIONS:
Drug: iv SPM 927 and oral placebo tablet — 60-minute infusion iv SPM 927 and oral placebo tablet
  Other Names: Lacosamide; Vimpat
  Arms: 1
Drug: oral SPM 927 tablet and iv placebo — 60-minute infusion placebo and oral SPM 927 tablet
  Other Names: Lacosamide; Vimpat
  Arms: 2
Drug: iv SPM 927 and oral placebo tablet — 30-minute infusion iv SPM 927 and oral placebo tablet
  Other Names: Lacosamide; Vimpat
  Arms: 3
Drug: oral SPM 927 tablet and iv placebo — 30-minute infusion placebo and oral SPM 927 tablet
  Other Names: Lacosamide; Vimpat
  Arms: 4

SUMMARY:
The purpose of this trial was to evaluate the safety and tolerability of SPM 927 when given as iv infusions compared with oral administration of the same dose strengths in subjects who were receiving oral SPM 927 for partial seizures with or without secondary generalization.

Trial procedures will include medical history update, physical/ neurological exams, ECGs, blood /urine sample collections and seizure diary completion.

Subjects completing the trial will return to the OLE trial to resume dosing with oral SPM 927.

ELIGIBILITY:
Inclusion Criteria:

* Subject with partial seizures with or without secondary generalization

Exclusion Criteria:

* Subject had previously received iv SPM 927
* Subject met the withdrawal criteria for the open-label extension trial with SPM 927 or was experiencing an ongoing serious adverse event.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2004-03-04 (Actual); Primary Completion 2004-08-17 (Actual); Study Completion 2004-11-30 (Actual)

PRIMARY OUTCOMES:
Adverse events, Vital signs, electrocardiograms,Physical examination, neurological examination | 2 Days

SECONDARY OUTCOMES:
Seizure counts | 2 days

CONTACTS AND LOCATIONS:
Overall Officials: UCB Clinical Trial Call Center, Study Director — +1 877 822 9493 (UCB)

REFERENCES:
- [Result] Biton V, Rosenfeld WE, Whitesides J, Fountain NB, Vaiciene N, Rudd GD. Intravenous lacosamide as replacement for oral lacosamide in patients with partial-onset seizures. Epilepsia. 2008 Mar;49(3):418-24. doi: 10.1111/j.1528-1167.2007.01317.x. Epub 2007 Sep 19. PMID 17888078
- See also: Clinical Study Summary on UCB.com — https://www.ucb.com/website/_up/ucb_com_patients/documents/SP616_CSS_20081118.pdf